CLINICAL TRIAL: NCT06736314
Title: A Single-center Exploratory Clinical Study on the Use of Removable Titanium Clips for the Treatment of Acute Variceal Hemorrhage from the Gastric Fundus
Brief Title: Removable Titanium Clip Treatment for Acute Variceal Hemorrhage from the Gastric Fundus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shupei Li (Other)
Responsible Party: Sponsor-Investigator, Shupei Li, student, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLLFS-24-26
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Gastric Variceal Bleeding
Keywords: a removable titanium clip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a removable titanium clip (Experimental)
  Interventions: Device: a removable titanium clip

INTERVENTIONS:
Device: a removable titanium clip — The removable titanium clip is a new type of titanium clip that offers advantages such as easy operation and convenient disassembly.

SUMMARY:
Removable Titanium Clip Treatment for Acute Variceal Hemorrhage from the Gastric Fundus

DETAILED DESCRIPTION:
During the procedure, a removable titanium clip was used to block the bleeding vessels, enabling rapid hemostasis. Five days later, secondary preventive measures such as ECI or TIPS were performed. The titanium clip was removed during or after the procedure, avoiding its retention in the body, which could interfere with subsequent MRI examinations and related treatments. In situations where emergency ECI or other treatments are not feasible, this method can serve as a 'temporary bridge' for the treatment of acute gastric fundal variceal hemorrhage, potentially saving the patient's life.

ELIGIBILITY:
Inclusion Criteria:

1. The patient and their family agree to and sign the relevant informed consent form.
2. Diagnosed with cirrhosis based on clinical manifestations, laboratory tests, imaging findings, or pathological examinations.
3. History of symptoms related to variceal upper gastrointestinal bleeding, such as hematemesis, melena, or rectal bleeding.
4. Patients confirmed by endoscopy to have bleeding from ruptured gastric varices.
5. Patients who are hemodynamically stable before or after initial fluid resuscitation.
6. Aged 18 to 75 years.

Exclusion Criteria:

1. Those with concomitant bleeding from ruptured esophageal varices.
2. A history of gastrointestinal-related surgical procedures.
3. Individuals with altered consciousness who are difficult to treat.
4. Those with concomitant malignant tumors.
5. Individuals with serious diseases involving the heart, brain, lungs, or kidneys.
6. Pregnant and breastfeeding women.
7. Those with contraindications to relevant treatments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate within 5 days after treatment | within 5 days after treatment
  Signs of rebleeding: A clinically significant event of active bleeding after hemostasis (hematemesis, melena, or rectal bleeding; a decrease in systolic blood pressure of >20 mmHg or an increase in heart rate of >20 beats/min; a drop in hemoglobin of >30 g/L without blood transfusion). (1) Early rebleeding: Occurs within 120 hours to 6 weeks after hemostasis. (2) Delayed rebleeding: Occurs more than 6 weeks after hemostasis. Non-EVB patients are excluded.

CONTACTS AND LOCATIONS:
Locations (1):
- Removable Titanium Clip, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No